CLINICAL TRIAL: NCT04740515
Title: Evaluation of the Influence of a Pharmacist-led Patient-Centered Medication Therapy Management on Adherence and Clinical Outcomes Among Preterm Infants With Iron Supplementation
Brief Title: Influence of a PPMTM on Adherence and Clinical Outcomes Among Preterm Infants With Iron Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaoxing Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Xu Renjie, Department of Clinical pharmacy, Shaoxing Maternity and Child Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XRenjie
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Preterm Infants; Clinical Outcome; Pharmaceutical Care
Keywords: Pharmaceutical Care; Medication Adherence; Iron Supplementation
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Involvement of pharmacists in improving medication (Experimental): Pharmacists involved care group. Tools used to improve medication adherence, (1)Patient medication guide (2)tailored Short Messaging Service (SMS) (3)Pharmaceutical follow-up
  Interventions: Other: pharmacists involved PPMTM
- usual care only (No Intervention): Patients were provided with usual care.

INTERVENTIONS:
Other: pharmacists involved PPMTM — This was an open labelled randomised study. Preterm Infants With iron supplementation were recruited and arbitrarily divided into the intervention group (usual care plus PPMTM) and the non-intervention group (usual care only). Those enrolled in the research were scheduled for follow-up for eight consecutive visits. Improvements in lab results and direct costs were compared longitudinally (pre and post analysis) between the groups.
  Arms: Involvement of pharmacists in improving medication

SUMMARY:
This is a randomised trial on the efficacy of a Pharmacist-led Patient-Centered Medication Therapy Management on clinical outcomes among preterm infants born before 32 weeks gestation with iron supplementation. The purpose of this study is to evaluate clinical outcome in the PPMTM program compared with usual care in an integrated health care system.

DETAILED DESCRIPTION:
This is a randomised trial on the efficacy of a Pharmacist-led Patient-Centered Medication Therapy Management on clinical outcomes among preterm infants born before 32 weeks gestation with iron supplementation. As a result, the Committee on Nutrition of the American Academy of Pediatrics (AAP) recommends daily oral iron supplementation, of at least 2-4 mg/kg/day from 2 weeks of age, to prevent iron deficiency in extremely premature infants. The purpose of this study is to evaluate clinical outcome in the PPMTM program compared with usual care in an integrated health care system.

ELIGIBILITY:
Inclusion Criteria:

* NICU inpatients between 26 and 32 weeks of gestation Infants older than two week of age and Iron dosing will be adjusted for weight at weekly intervals to maintain dosing at 4mg/kg/day.

Parental permission obtained prior to start of study

Exclusion Criteria:

* In extremis during consent window (as judged by primary attending provider) Known or suspected genetic disorder Small for gestational age (birth weight below the 10th percentile for gestational age) Unable to return for follow-up evaluation at 6 months of age

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
ferritin level | At discharge or 40 weeks corrected age (whichever occurs first), Correct gestational age of 3 months and 6 months
  Iron insufficiency will be determined by ferritin level less than 70 ng/mL
hemoglobin level | At discharge or 40 weeks corrected age (whichever occurs first), Correct gestational age of 3 months and 6 months
  Iron insufficiency will be determined by hemoglobin level less than 8 g/dL
reticulocyte hemoglobin equivalent (Ret-He, pg) | At discharge or 40 weeks corrected age (whichever occurs first), Correct gestational age of 3 months and 6 months
  Iron insufficiency will be determined by Ret-He less than 27.2 pg
reticulocyte count (%) | At discharge or 40 weeks corrected age (whichever occurs first), Correct gestational age of 3 months and 6 months
  Iron insufficiency will be determined by reticulocyte count less than 2%

CONTACTS AND LOCATIONS:
Overall Officials: Renjie Xu, PhD, Principal Investigator — Shaoxing Maternity and Child Health Care Hospital
Locations (1):
- Shaoxing Maternity and Child Care hospital, Shaoxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided